CLINICAL TRIAL: NCT00453713
Title: Determinants of Outcome in Diffuse Parenchymal Lung Disease
Brief Title: Race, Ethnicity, and Diffuse Parenchymal Lung Disease
Status: Completed | Type: Observational
Sponsor: Columbia University (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, David J. Lederer, M.D., Irving Assistant Professor of Medicine (in Pediatrics), Columbia University
Other Study IDs: AAAB8771; K23HL086714 (NIH)
Record Dates: First submitted 2007-03-27; First posted 2007-03-29 (Estimated); Last update posted 2015-04-21 (Estimated); Status verified 2015-04

CONDITIONS: Idiopathic Pulmonary Fibrosis; Interstitial Lung Disease; Diffuse Parenchymal Lung Disease
Keywords: Idiopathic pulmonary fibrosis; Interstitial lung disease; Diffuse parenchymal lung disease; Health disparities
MeSH Terms: conditions — Idiopathic Pulmonary Fibrosis; Lung Diseases, Interstitial

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Plasma/serum, DNA, and circulating cells and endothelial microparticles will be collected and processed.
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to identify factors that contribute to higher mortality rates among blacks and Hispanics with diffuse parenchymal lung disease.

DETAILED DESCRIPTION:
It is well known that both socioeconomic and biological factors may contribute to race- and ethnicity-based health disparities. Black and Hispanic Americans have worse access to healthcare services and tend to receive care from physicians who cannot themselves access the same services for their patients that physicians who care for white patients can. These factors may play important roles in the development and maintenance of health disparities. In addition, biological differences may contribute to disparities. We propose to identify factors that explain survival disparities in a group of lung diseases called diffuse parenchymal lung diseases (DPLDs), including a severe form of DPLD called idiopathic pulmonary fibrosis (IPF). We will follow patients with DPLD at our center and measure both social and biological factors to try to identify the factors that lead to survival disparities between races. Results of this study will be used to design clinical trials aimed at reducing these disparities.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of IPF or other DPLD according to ATS criteria
* Signed informed consent

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Diffuse parenchymal lung disease
Sampling Method: Non-Probability Sample
Enrollment: 565 (Actual)
Dates: Start 2006-07; Primary Completion 2013-08 (Actual); Study Completion 2013-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David J Lederer, M.D., Principal Investigator — Columbia University
Locations (1):
- Columbia University Medical Center, New York, New York, United States